CLINICAL TRIAL: NCT01159249
Title: A Multicenter, Open Label, Long-Term Safety Study of 52 Weeks Treatment With Vildagliptin in Patients With Type 2 Diabetes
Brief Title: Long-term Safety Study of Vildagliptin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237A1308
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2012-05

CONDITIONS: Type 2 Diabetes
Keywords: Vildagliptin, Type 2 Diabetes, HbA1c, Fasting Plasma Glucose, Long-Term Safety
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

ARMS (4):
- Open Met add-on vildagliptin (Other)
  Interventions: Drug: Vildagliptin
- Open TZD add-on vildagliptin (Other)
  Interventions: Drug: Vildagliptin
- Open α-GI add-on vildagliptin (Other)
  Interventions: Drug: Vildagliptin
- Glinides add-on vildagliptin (Other)
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
This study is designed to demonstrate the long-term safety of vildagliptin in patients with type 2 diabetes. This study will study vildagliptin as add-on therapy with metformin, thiazolidinedione, α-glucosidase inhibitor (α-GI), rapid-acting insulin secretagogues in the treatment of type 2 diabetes in Japan.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes inadequately controlled with diet, exercise and metformin, thiazolidinedione, or α-GI, or glinides monotherapy
* Age in the 20 years or over inclusive
* HbA1c in the range of ≥ 6.5 to ≤ 10%

Exclusion Criteria:

* Type 1 diabetes mellitus, diabetes that is a result of pancreatic injury, or secondary forms of diabetes
* Significant heart diseases
* Significant diabetic complications

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Measure AEs, vital signs, laboratory evaluations | 52 weeks

SECONDARY OUTCOMES:
HBA1c | 52 weeks
Fasting Plasma Glucose | 52 weeks
Fasting Insulin | 52 weeks
Fasting C-peptide | 52 weeks
HOMA-B | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals Corporation, Study Director — Novartis Pharmaceuticals
Locations (20):
- Japan (20):
  - Novartis Investigative Site, Hunabashi, Chiba
  - Novartis Investigative Site, Chikushino-shi, Fukuoka
  - Novartis Investigative Site, Itoshima-shi, Fukuoka
  - Novartis Investigative Site, Kōriyama, Fukushima
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Izumisano, Osaka
  - Novartis Investigative Site, Hannou, Saitama
  - Novartis Investigative Site, Hiki-Gun, Saitama
  - Novartis Investigative Site, Kawaguchi, Saitama
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Edogawa-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Katsushika-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
  - Novartis Investigative Site, Fukuoka

REFERENCES:
- See also: Results for CLAF237A1308 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7543